CLINICAL TRIAL: NCT05865132
Title: CDK4/6 Inhibitor Palbociclib Combined With Afatinib as Second-line Treatment for Advanced Squamous Carcinoma of the Esophagus or Gastroesophageal Junction Progressed on at Least First-line Chemotherapy: a Phase 2 Trial
Brief Title: Palbociclib Combined With Afatinib for Advanced Squamous Carcinoma of Esophagus or Gastroesophageal Junction
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AIPING ZHOU (Other)
Responsible Party: Sponsor-Investigator, AIPING ZHOU, Vice director of Department of Medical Oncology, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC3628
Record Dates: First submitted 2023-04-11; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Esophagus Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — palbociclib; Afatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Palbociclib + Afatinib (Experimental): The first 6 enrolled patients were treated with Palbociclib 125 mg po qd on day 1 to 21, Afatinib 40 mg po qd on day 1 to 14, every 28 days as a cycle; If there are ≥ 2 cases of dose-limiting toxicity (DLT), the following 6 patients will reduce the dose to Palbociclib 125mg po qd on day 1 to 21, Afatinib 30mg po qd on day 1 to 28, every 28 days as a cycle; If ≥ 2 cases of DLT occur again, the following 6 patients will reduce the dose to Palbociclib 100mg po qd on day 1 to 21, Afatinib 30mg po qd on day 1 to 28, every 28 days as a cycle; If ≥ 2 cases of DLT occur again, we will analyze the characteristics of adverse events and determine the subsequent dose.
  Interventions: Drug: Palbociclib; Drug: Afatinib

INTERVENTIONS:
Drug: Palbociclib — 120mg/125mg po qd on day 1 to 21, every 28 days
Drug: Afatinib — 30mg/40mg po qd on day 1 to 28, every 28 days

SUMMARY:
This is a prospective, multicenter, exploratory study. Patients with advanced esophageal or gastro-esophageal junction squamous carcinoma who had progressed on first-line chemotherapy combined with immune checkpoint inhibitors were treated with CDK4/6 inhibitor Palbociclib combined with Afatinib. Dose titration was used to determine the final dose, and objective antitumor efficacy was evaluated every 2 cycles (8 weeks +/- 7 days) according to RECIST 1.1 criteria, until tumor progression, intolerable toxicity, death, or withdrawal of informed consent. The primary endpoint is the objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed metastatic or inoperable locally advanced squamous carcinoma of the esophagus or gastroesophageal junction that is not amenable to radical radiotherapy.
* Prior progression to at least first-line chemotherapy which must include immune checkpoint inhibitors (except in patients with contraindications to immune checkpoint inhibitors). Adjuvant/neoadjuvant therapy is allowed and is considered first-line therapy for advanced disease if recurrence occurs during or within 6 months of completion of adjuvant/neoadjuvant therapy.
* At least one measurable tumor lesion according to RECIST V1.1 criteria. A lesion previously treated with radiotherapy is not acceptable as a target lesion unless the lesion is significantly progressive.
* Sign the informed consent form
* 18~75 years
* Performance status: ECOG 0-1
* Good organ function:

Blood routine: hemoglobin ≥90g/L, neutrophil ≥1.5×10^9/L, platelet ≥100×10^9/L; Renal function: creatinine≤1.5×upper limit of normal (UNL) or creatinine clearance ≥50ml/min; Liver function: total bilirubin (TBIL)≤1.5×upper limit of normal (UNL); ALT≤2.5×UNL, AST≤2.5×UNL; Ejection fraction at least 50% (or lower limit of normal) by echocardiogram

Exclusion Criteria:

* Other pathological category, such as adenocarcinoma, adenosquamous carcinoma
* Have received CDK4/6 inhibitors or anti-EGFR targeted drugs in the past
* Known to have allergic reactions to any ingredients or excipients of experimental drugs
* Unable to swallow or under other circumstance which would drug absorption
* Other active malignant tumors, excluding those who have been disease free for more than 5 years or in situ cancer considered to have been cured by adequate treatment
* Diabetes was not controlled, defined as HbA1c > 7.5% after anti-diabetic drugs or hypertension was not controlled, defined as systolic / diastolic blood pressure > 140 / 90 mmHg after antihypertensive drug
* Myocardial infarction, severe/unstable angina, New York Heart Association (NYHA) class III or IV congestive heart failure in the past 12 months
* Known to be infected with human immunodeficiency virus (HIV), have acquired immunodeficiency syndrome (AIDS) related diseases, have active hepatitis B or hepatitis C
* Pregnant or nursing
* May increase the risk associated with participation in the study or administration of the study drug or mental illness that may interfere with the interpretation of research results
* There are other serious diseases that the researchers believe patients cannot be included in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
ORR | 3 years
  objective response rate

SECONDARY OUTCOMES:
DCR | 3 years
  disease control rate
PFS | From date of initiation of treatment to date of progression or death due to any cause, whichever occurs first up to 3 years
  progression free survival
OS | From date of initiation of treatment to date of death up to 3 years
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided